CLINICAL TRIAL: NCT00724464
Title: A Greek Observational Study on Relapse Rate and Sustained Virological Response in Naive CHC Patients, Treated With Pegylated Interferon Alpha-2b and Ribavirin in Daily Clinical Practice
Brief Title: Efficacy of PegIntron (Peginterferon Alfa-2b) and Rebetol (Ribavirin) in Treatment-naïve Subjects With Chronic Hepatitis C in Clinical Practice in Greece (Study P05209)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P05209
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Results first posted 2011-11-08 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Hepatitis C, Chronic; Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with Chronic Hepatitis C: Treatment-naïve participants with chronic hepatitis C, undergoing treatment with a standard treatment regimen of PegIntron and Rebetol in clinical practice at approximately 28 sites in Greece
  Interventions: Biological: PegIntron (peginterferon alfa-2b, pegylated interferon alfa-2b); Drug: Rebetol (ribavirin)

INTERVENTIONS:
Biological: PegIntron (peginterferon alfa-2b, pegylated interferon alfa-2b) — Prior to enrollment in the study, PegIntron was to be administered at a dose of 1.5 μg/kg/week subcutaneously in accordance with approved labeling. Therapy duration varied from 24 to 48 weeks depending on HCV viral load and genotype followed by a 24-week post-treatment follow-up.
  Other Names: SCH 54031
Drug: Rebetol (ribavirin) — Prior to enrollment in the study, Rebetol was to be administered at a dose of 800-1200 mg/day orally in accordance with approved labeling. Therapy duration varied from 24 to 48 weeks depending on HCV viral load and genotype followed by a 24-week post-treatment follow-up.
  Other Names: SCH 18908

SUMMARY:
The objective of the study is to evaluate the rates of Hepatitis C virus (HCV) eradication and relapse in participants treated with PegIntron and Rebetol in clinical practice in Greece. Participants will not be treated as part of the study. Data on participants treated in accordance with approved labeling will be collected retrospectively from approximately 30 sites in Greece.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have already begun Summary of Product Characteristics (SmPC)-based combination treatment with pegylated interferon alpha-2b and ribavirin, prior to the site initiation date.
* Participants who have been receiving combination treatment with pegylated interferon alpha-2b and ribavirin for at least 6 months before enrollment.
* Participants who have achieved negative HCV RNA at the end of treatment, defined according to genotype (24 weeks for HCV genotypes 2/3 and 48 weeks for genotypes 1/4).
* Participants with diagnosed chronic hepatitis C (CHC) and HCV genotype 1, 2, 3 or 4.
* Participants older than 18 years, regardless of gender or race.

Exclusion Criteria:

* The participant has received treatment for CHC in the past (not treatment-naive).
* The participant has received treatment in the context of a clinical trial in the participating site.
* The participant has been diagnosed with a concomitant infection e.g. with hepatitis B or HIV
* The participant has de-compensated liver disease or belongs to a special population, such as liver transplant, hemophilia, severe pre-existing psychiatric disorder, auto-immune disease, thalassaemia.
* The participant has positive HCV RNA at the end of treatment.
* Pregnant women or women intending to bear children or sexual partners of women wishing to bear children and for a 7-month period after the end of treatment, as indicated in the SmPC of Rebetol.
* The participant is not eligible on grounds of contra-indications, special warnings, particular population and/or the section on pregnancy and lactation of the SmPC.
* The participant has interrupted treatment for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Treatment-naïve participants with chronic hepatitis C treated with PegIntron and Rebetol in accordance with approved labeling in clinical practice in Greece prior to enrollment in the current study. Data from patients treated at approximately 28 sites will be retrospectively analyzed.
Sampling Method: Probability Sample
Enrollment: 332 (Actual)
Dates: Start 2007-12; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 401 participants were screened for eligibility. 332 participants were enrolled in the study.
Groups:
- Pegylated Interferon Alpha-2b and Ribavirin: Participants with CHC of any genotype were treated with a standard treatment regimen of pegylated interferon alfa-2b and ribavirin. Each dose of pegylated interferon alfa-2b was administered as a subcutaneous injection calculated as 1.5 μg/kg once a week. Ribavirin was taken orally, twice daily, at a daily dose of 800 to 1200 mg. Therapy duration varied from 24 to 48 weeks depending on HCV genotype and viral load followed by a 24-week post-treatment follow-up.
Period: Overall Study
Arm/Group | Pegylated Interferon Alpha-2b and Ribavirin
Started | 332
Completed | 309
Not Completed | 23

BASELINE CHARACTERISTICS:
Arm/Group | Pegylated Interferon Alpha-2b and Ribavirin
Number analyzed (Participants) | 332
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102
  Male | 230

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved Sustained Virological Response as Assessed at 24-week Post-treatment Follow-up
Description: Sustained virological response (SVR) was assessed at the 24-week post-treatment follow-up (Visit 2). SVR was defined as undetectable plasma Hepatitis C virus Ribonucleic acid (HCV-RNA) at 24 weeks after termination of combination treatment (24 or 48 weeks of treatment duration).
Time Frame: 24 weeks following completion of 24 or 48 weeks of therapy
Population: Efficacy Analysis Set (EAS) included all participants enrolled into the study who attended the final study visit and had HCV RNA evaluation measurement available at the 24-week post-treatment follow-up.
Measure: Number; unit: Participants
Groups:
- Pegylated Interferon Alpha-2b and Ribavirin: Participants with Chronic Hepatitis C (CHC) of any genotype were treated with a standard treatment regimen of pegylated interferon alfa-2b and ribavirin. Each dose of pegylated interferon alfa-2b was administered as a subcutaneous injection calculated as 1.5 μg/kg once a week. Ribavirin was taken orally, twice daily, at a daily dose of 800 to 1200 mg. Therapy duration varied from 24 to 48 weeks depending on Hepatitis C virus (HCV) genotype and viral load followed by a 24-week post-treatment follow-up.
Arm/Group | Pegylated Interferon Alpha-2b and Ribavirin
Number analyzed (Participants) | 309
Participants | 286

2. Secondary Outcome: Number of Participants Who Achieved Sustained Virological Response as Assessed at 24-week Post-treatment Follow-up by Subgroups Based on HCV Genotype at Baseline
Description: SVR was assessed at the 24-week post-treatment follow-up (Visit 2) by subgroups based on HCV genotype (1, 2, 3, 4, or 2 & 3) at baseline. SVR was defined as undetectable plasma HCV-RNA at 24 weeks after termination of combination treatment (24 or 48 weeks of treatment duration).
Time Frame: 24 weeks following completion of 24 or 48 weeks of therapy
Population: Efficacy Analysis Set (N=309) included all participants enrolled into the study who attended the final study visit and had HCV RNA evaluation measurement available at the 24-week post-treatment follow-up. Of the 309 participants in this population, 286 achieved SVR and were included in this analysis. 23 participants were relapsers.
Measure: Number; unit: Participants
Arm/Group | Pegylated Interferon Alpha-2b and Ribavirin
Number analyzed (Participants) | 286
Participants
  Genotype 1 | 81
  Genotype 2 | 28
  Genotype 3 | 146
  Genotype 4 | 30
  Genotype 2 & 3 | 1

3. Primary Outcome: Number of Participants Who Demonstrated Virological Relapse as Assessed at 24-week Post-treatment Follow-up
Description: Virological relapse was assessed at the 24-week post-treatment follow-up (Visit 2). Virological relapse was defined as undetectable plasma HCV-RNA at end of combination treatment (Visit 1- considered Week 24 or Week 48 after treatment start depending on treatment duration), but with positive HCV-RNA at the 24-week post treatment follow-up.
Time Frame: 24 weeks following completion of 24 or 48 weeks of therapy
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Pegylated Interferon Alpha-2b and Ribavirin
Number analyzed (Participants) | 309
Participants | 23

4. Secondary Outcome: Number of Participants Who Achieved Sustained Virological Response as Assessed at 24-week Post-treatment Follow-up by Subgroups Based on Liver Fibrosis Stage at Baseline
Description: SVR was assessed at the 24-week post-treatment follow-up (Visit 2) by subgroups based on liver fibrosis stage, where biopsy was available, at baseline: absence, minimal, moderate, or significant as assessed by investigator. SVR was defined as undetectable plasma HCV-RNA at 24 weeks after termination of combination treatment (24 or 48 weeks of treatment duration).
Time Frame: 24 weeks following completion of 24 or 48 weeks of therapy
Population: Efficacy Analysis Set (N=309) included all participants enrolled into the study who attended the final study visit and had HCV RNA evaluation measurement available at the 24-week post-treatment follow-up. Of the 309 participants in this population, 286 achieved SVR and were included in this analysis. There was missing data for 157 participants.
Measure: Number; unit: Participants
Arm/Group | Pegylated Interferon Alpha-2b and Ribavirin
Number analyzed (Participants) | 286
Participants
  Absence | 83
  Minimal | 27
  Moderate | 15
  Significant | 4
  Missing | 157

5. Secondary Outcome: Number of Participants Who Achieved Sustained Virological Response as Assessed at 24-week Post-treatment Follow-up by Subgroups Based on HCV-RNA Viral Load at Baseline
Description: SVR was assessed at the 24-week post-treatment follow-up (Visit 2) by subgroups based on HCV-RNA viral load at baseline as assessed by investigator. Low viral load was defined as <400,000 International Units/milliliter (IU/mL) and high viral load was defined as >=400,000 IU/mL. SVR was defined as undetectable plasma HCV-RNA at 24 weeks after termination of combination treatment (24 or 48 weeks of treatment duration).
Time Frame: 24 weeks following completion of 24 or 48 weeks of therapy
Population: Efficacy Analysis Set (N=309) included all participants enrolled into the study who attended the final study visit and had HCV RNA evaluation measurement available at the 24-week post-treatment follow-up. Of the 309 participants in this population, 286 achieved SVR and were included in this analysis. There was missing data for 32 participants.
Measure: Number; unit: Participants
Arm/Group | Pegylated Interferon Alpha-2b and Ribavirin
Number analyzed (Participants) | 286
Participants
  Low Viral Load | 99
  High Viral Load | 155
  Missing | 32

6. Secondary Outcome: Number of Participants Who Achieved Sustained Virological Response as Assessed at 24-week Post-treatment Follow-up by Subgroups Based on Alanine Aminotransferase (ALT) Levels at Baseline
Description: SVR was assessed at the 24-week post-treatment follow-up (Visit 2) by subgroups based on ALT levels at baseline as assessed by investigator. Normal baseline ALT level was defined as <40 IU/mL and elevated baseline ALT level was defined as >= 40 IU/mL. SVR was defined as undetectable plasma HCV-RNA at 24 weeks after termination of combination treatment (24 or 48 weeks of treatment duration).
Time Frame: 24 weeks following completion of 24 or 48 weeks of therapy
Population: Efficacy Analysis Set (N=309) included all participants enrolled into the study who attended the final study visit and had HCV RNA evaluation measurement available at the 24-week post-treatment follow-up. Of the 309 participants in this population, 286 achieved SVR and were included in this analysis. There was missing data for 6 participants.
Measure: Number; unit: Participants
Arm/Group | Pegylated Interferon Alpha-2b and Ribavirin
Number analyzed (Participants) | 286
Participants
  Normal Baseline ALT levels | 28
  Elevated Baseline ALT levels | 252
  Missing | 6

7. Secondary Outcome: Number of Participants Who Achieved Sustained Virological Response as Assessed at 24-week Post-treatment Follow-up by Subgroups Based on Study Treatment Dosage Modification
Description: SVR was assessed at the 24-week post-treatment follow-up (Visit 2) by subgroups based on study treatment dosage modification: no dosage modification or any dosage modification of study treatment. SVR was defined as undetectable plasma HCV-RNA at 24 weeks after termination of combination treatment (24 or 48 weeks of treatment duration).
Time Frame: 24 weeks following completion of 24 or 48 weeks of therapy
Population: Efficacy Analysis Set (N=309) included all participants enrolled into the study who attended the final study visit and had HCV RNA evaluation measurement available at the 24-week post-treatment follow-up. Of the 309 participants in this population, 286 achieved SVR and were included in this analysis.
Measure: Number; unit: Participants
Arm/Group | Pegylated Interferon Alpha-2b and Ribavirin
Number analyzed (Participants) | 286
Participants
  No Dosage Modification of Study Treatment | 234
  Any Dosage Modification of Study Treatment | 52

8. Secondary Outcome: Number of Participants Who Achieved Sustained Virological Response as Assessed at 24-week Post-treatment Follow-up by Subgroups Based on Achievement of Rapid Virological Response
Description: SVR was assessed at the 24-week post-treatment follow-up (Visit 2) by subgroups based on achievement of rapid virological response (RVR) where data was available. RVR was defined as negative HCV-RNA after 4 (+/- 1) weeks of treatment. SVR was defined as undetectable plasma HCV-RNA at 24 weeks after termination of combination treatment (24 or 48 weeks of treatment duration).
Time Frame: 24 weeks following completion of 24 or 48 weeks of therapy
Population: Efficacy Analysis Set (N=309) included all participants enrolled into the study who attended the final study visit and had HCV RNA evaluation measurement available at the 24-week post-treatment follow-up. Of the 309 participants in this population, 286 achieved SVR and were included in this analysis. There was missing data for 250 participants.
Measure: Number; unit: Participants
Arm/Group | Pegylated Interferon Alpha-2b and Ribavirin
Number analyzed (Participants) | 286
Participants
  RVR at Week 4 (+/- 1) | 20
  Non-RVR at Week 4 (+/- 1) | 16
  Missing | 250

9. Secondary Outcome: Number of Participants Who Achieved Sustained Virological Response as Assessed at 24-week Post-treatment Follow-up by Subgroups Based on Compliance With the 80/80/80 Rule
Description: SVR was assessed by subgroups based on compliance with the 80/80/80 rule where data was available. 80/80/80 compliant participants were those that received >= 80% of the planned total doses of both pegylated interferon alfa-2b & ribavirin for >=80% of the duration of therapy. 3 rates were to be computed: Compliance with study duration, compliance with pegylated interferon dose, & compliance with ribavirin dose. A participant was defined as compliant, if none of the 3 rates were < than 80%. SVR was defined as undetectable plasma HCV-RNA at 24 weeks after termination of combination treatment.
Time Frame: 24 weeks following completion of 24 or 48 weeks of therapy
Population: No data had been captured in the Case Report Forms, and therefore no relevant analysis had been performed.
Arm/Group | Pegylated Interferon Alpha-2b and Ribavirin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The safety population included the total number of participants screened for eligibility (N=401). This population includes the total number of eligible participants enrolled in the study or the Full Analysis Set (N=332) and the non-eligible participants or the screening failure set (N=69).
Arm/Group | Pegylated Interferon Alpha-2b and Ribavirin
Serious Adverse Events (participants affected / at risk) | 5/401
Other Adverse Events (participants affected / at risk) | 123/401
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegylated Interferon Alpha-2b and Ribavirin (N=401)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Lung Infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Tooth Abscess (Infections and infestations) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Emotional Disorder (Psychiatric disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegylated Interferon Alpha-2b and Ribavirin (N=401)
Anaemia (Blood and lymphatic system disorders) | 61 (61)
Leukopenia (Blood and lymphatic system disorders) | 31 (32)
Fatigue (General disorders) | 38 (41) — Includes Fatigue, Lassitude, and Fatigability
Weight Decreased (Investigations) | 27 (27)
Alopecia (Skin and subcutaneous tissue disorders) | 21 (21) — Includes Alopecia, Hair Loss, and Accelerated Hair Loss

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The principal investigator agrees not to publish or publicly present any interim results of the Study without prior written consent of the SPONSOR. The principal investigator further agrees to provide forty-five (45) days written notice to the SPONSOR prior to submission for publication or presentation

to permit the SPONSOR to review copies of abstracts or manuscripts for publication which report any results of the Study. The SPONSOR shall have the right to review & comment on any presentation.